CLINICAL TRIAL: NCT02368808
Title: Coping With Loss: A Bereavement Initiative for Adolescent Girls in the Free State, South Africa
Brief Title: Adolescent Bereavement Initiative in the Free State, South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University School of Social Work (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Tonya Renee Thurman, Associate Professor, Tulane University School of Social Work
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AID-674-A-12-00002-CWL
Record Dates: First submitted 2015-02-09; First posted 2015-02-23 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Grief; Bereavement
Keywords: orphans and vulnerable children; South Africa; peer support group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abangane Support Group (Experimental): Bereavement support group for adolescents
  Interventions: Behavioral: Abangane Support Group
- Wait List (No Intervention): Wait-listed adolescents will be able to participate in Abangane at the close of the study.

INTERVENTIONS:
Behavioral: Abangane Support Group — The Abangane support group program consists of 8 sessions for bereaved adolescents with standardized activities and discussion content based the Khululeka Grief Support Program in Cape Town, South Africa. The materials include a resource book that provides training and referral agencies for grief group facilitators as well as exercises and creative activities designed to stimulate group discussions that will help adolescents to deal with loss and grief.
  Arms: Abangane Support Group

SUMMARY:
Coping with Loss is a randomized controlled trial to assess the effectiveness of a bereavement intervention targeting female adolescents who have experienced the death of someone important in their lives. Adolescents aged 12 and older in the Free State province of South Africa will be invited to participate in an 8-session school-based peer support group focused on coping with loss. Interventions will be implemented by Social Workers from Child Welfare Bloemfontein and Childline Free State (CWBFN & CLFS) that have provided support services for orphans and vulnerable children (OVC) in the Free State Province since 2013. The study population will be identified through the CWBFN & CLFS intake process and consist of bereaved female adolescents from up to 11 participating schools. Eligible adolescents will be randomly assigned to receive the intervention in 2015 or wait-listed for enrollment following the study period. Survey data will be collected from adolescents and caregivers before and two months following the completion of the interventions. Data will be analyzed to assess for pre- and post-test differences between the intervention and wait-listed group on key psychosocial outcomes, including measures of grief, resilience, mental health, social support, academic competence and adolescent-caregiver interactions.

DETAILED DESCRIPTION:
The HIV/AIDS epidemic, accidental injuries and violence have gradually increased the mortality rate among prime age adults in South Africa since 1997 (Statistics South Africa, 2006) leading to an increase in the number of children experiencing bereavement. Of the approximately four million orphans in South Africa in 2012, over half (62.5%) are due to parental death from AIDS (UNICEF, 2013). Studies have found that parental loss in childhood and adolescence is associated with a range of immediate and later life outcomes including problems at school, depression, criminality, early sexual activity, and unemployment (Aynsley-Green, 2012). However, support counselling for bereaved children and adolescents is virtually nonexistent in South Africa (Collingwood, 2014) and children are often not encouraged to express grief or participate in mourning rituals for the deceased. A randomized controlled trial of AIDS orphans in Uganda found that school-based peer support groups reduced the symptoms of anxiety, depression and anger compared to a control group that did not participate in the peer support groups (Kumakech, 2009). This base of evidence demonstrates both the unmet need and potential impact of a bereavement initiative that will be offered by CWBFN & CLFS in Free State. This research will contribute to the evidence base for effective programming for bereaved adolescents in South Africa as well as other high HIV prevalence populations.

The aim of this study is to assess the effectiveness of time-limited adolescent grief counseling peer groups in improving the psychosocial wellbeing of bereaved female adolescents. Results from the study will be used to develop evidence-based youth bereavement counselling programs to be implemented in additional areas of South Africa. The results will be presented to South African OVC social service organizations as well as submitted to peer-reviewed scientific journals for wider dissemination.

(Note that the original study design included a family component/sessions for caregivers that was not able to be realized by the program implementers)

ELIGIBILITY:
Inclusion Criteria:

* Attends one of the participating schools
* English or Sesotho speaker

Exclusion Criteria:

* Previous participation in CWBFN&CLFS grief counselling group

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 843 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in Grief Intensity | Baseline, 2 months post-intervention
  Grief intensity, including general grief, intrusive thoughts and prolonged grief, is assessed through adolescent self-report of items from three standardized scales (1) Core Bereavement Items (CBI) five-item grief subscale (Burnett et al, 1997); (2) Intrusive Grief Thoughts Scale (IGTS) (ASU Program for Prevention Research, 1999); and the (3) Inventory of Complicated Grief -Revised for Children (ICG-RC) six-item screening tool (Melhem, Porta, Payne & Brent, 2013).
Change in Mental Health | Baseline, 2 months post-intervention
  Depressive symptomology will be assessed through adolescent self-report of the 20-item Center for Epidemiologic Studies Depression Scale for Children (CES-DC) (Weissman 1980, Faulstich 1986). Items assess the frequency of symptoms of depression including feelings of happiness, appetite, self-esteem, energy levels, sleep patterns, etc. Adolescent behaviour is assessed using the Brief Problem Monitor-Parent Form (BPM-P) (Achenbach 2011). BPM-P is a 19-item subset of the Child Behavior Checklist (CBCL) that captures problem behaviour, including internalizing and externalizing behaviour in children ages 6-18. Caregivers report on adolescent behaviour over the past four weeks.

SECONDARY OUTCOMES:
Change in Caregiver-Adolescent Interactions | Baseline, 2 months post-intervention
  Caregiver-Adolescent interactions are assessed through adolescent report of connectedness to caregiver and caregiver report of positive parenting practices, such as discipline, supervision, and supportiveness. Connectedness to Caregiver is assessed using the Inventory of Parent and Peer Attachment (Amsden & Greenberg, 1987). Positive parenting, discipline and supervision were measured using the Alabama Parenting Questionnaire short form (APQ-9) (Elgar et al). Harsh punishment is assessed through both caregiver and adolescent report using an adapted version of the Parent-Child Conflict Tactics Scale (CTSPC)'s psychological aggression and physical assault subscales (Straus et al., 1998). Supportiveness was measured with The Parent Behavior Inventory (PBI)'s Supportive/Engaged subscale, which measures parental affect towards the adolescent in their care (Lovejoy, Weis, O'hare & Rubin, 1999).
Change in Social Support | Baseline, 2 months post-intervention
  Social Support is assessed through items focused on social support received in dealing with the bereavement itself, basic social support, and emotional social support. Social support for coping with bereavement was measured using self-generated items, such as You can discuss your feelings about this loss with your family. Emotional social support is measured with the giving and receiving emotional support subscales of the 2-Way Social Support Scale (Shakespeare-Finch & Obst, 2011). Basic social support consists of four items from the MEASURE evaluation (Measure Evaluation, 2014).
Change in Academic Competence | Baseline, 2 months post-intervention
  Academic competence is assessed through adolescent self-report of academic self-efficacy, motivation and attendance. Academic self-efficacy is based on the academic self-efficacy subscale of the Self-Efficacy Questionnaire for Children (SEQ-C) (Muris, 2001) and assesses perceived performance in school including success in paying attention, passing tests, and completing homework. Academic motivation assesses the perceived importance of education and efforts to do well in school. Attendance is measured with one self-generated item which asks about absenteeism in the seven days prior to the survey, not including school holidays.
Change in Resilience | Baseline, 2 months post-intervention
  Resilience is assessed through positive appraisal coping abilities, including perceived coping, personal growth, emotional regulation and future expectations. Perceived coping is assessed with a self-generated scale based on items from the Grief Evaluation Measure (GEM) (Jordan & Baker, 2005). Personal growth as a result of the loss is assessed using the personal growth subscale of the Hogan Grief Reaction Checklist (Hogan, Greenfield & Schmidt, 2001). Emotional regulation is based on the adolescent's emotional self-efficacy, or perceived ability to regulate feelings and emotions, and is assessed with the emotional self-efficacy subscale of the Self-Efficacy Questionnaire for Children (SEQ-C) (Muris, 2001). Future expectations, or hopes for the future, is based on items from a self-generated scale used in a previous study of OVC in South Africa by the authors (Thurman, 2011) and an adapted subscale of the Social and Health Assessment (SAHA) (Ruchkin 2004).

CONTACTS AND LOCATIONS:
Overall Officials: Tonya R Thurman, MPH, PhD, Principal Investigator — Tulane University School of Social Work

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thurman TR, Luckett BG, Nice J, Spyrelis A, Taylor TM. Effect of a bereavement support group on female adolescents' psychological health: a randomised controlled trial in South Africa. Lancet Glob Health. 2017 Jun;5(6):e604-e614. doi: 10.1016/S2214-109X(17)30146-8. Epub 2017 Apr 24. PMID 28462880